CLINICAL TRIAL: NCT02333955
Title: A Phase 2 Extension of Study GCS-100-CS-4003
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCS-100-CS-4004
Record Dates: First submitted 2014-12-15; First posted 2015-01-08 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — GCS-100; citrus pectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 mg IV push (Experimental): GCS-100
  Interventions: Drug: GCS-100

INTERVENTIONS:
Drug: GCS-100 — 3 mg GCS-100 IV push. All doses of study drug will be administered least once monthly for a total of 1 year with a follow-up 4 weeks after the last dose is administered.
  Other Names: MCP (modified citrus pectin)

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of extended dosing with a fixed dose of GCS-100 3 mg IV push in patients with Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
Galectin-3 contributes to fibrosis, is elevated in patients with ESRD, and correlates with adverse outcomes (de Boer et. al., 2011, Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). Animal models with genetic knockout of galectin-3 demonstrate a reduction in structural and functional deficits in the kidney (Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). GCS-100 is a galectin-3 antagonist that has been shown to reduce fibrosis pre-clinically. Based on the role of galectin-3 and fibrosis in kidney disease, the Sponsor believes GCS-100 may be effective at treating patients with CKD.

This study will consist of a fixed dose of GCS-100 3mg IV push at least every 30 days for a total of 1 year with a follow-up 4 weeks after the last dose is administered.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of understanding the purpose and risks of the study and is able to provide written informed consent
2. Subject was enrolled in GCS-100-CS-4003.

Exclusion Criteria:

1. Subject experienced a Grade 3 or worse adverse event related to GCS-100 in clinical study GCS-100-CS-4003.
2. Systolic blood pressure ≤90 mmHg and ≥160 mmHg and diastolic blood pressure ≤40 mmHg and ≥100 mmHg at screening
3. Subject has clinical laboratory values of:

   * Hemoglobin: ≤9 g/dL
   * Total bilirubin: >1.5X the upper limit of normal (ULN)
   * ALT and/or AST: >2.5X ULN
4. Subject has a concomitant disease or condition, including laboratory abnormalities, which, in the opinion of the investigator, could interfere with the conduct of the study or put the subject at unacceptable risk.
5. Subject who may require renal replacement therapy within the next 2 months, at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and tolerability of extended dosing with a fixed dose of GCS-100 3 mg IV push in patients with CKD (side effects) | Participants will be followed for the duration of the study, up to 1 year with a four week additional follow-up period
  Evaluate side effects of this therapy when administered for an extended period of time. Determine response to therapy (by measuring kidney function monthly) as compared to subjects' response in study GCS-100-CS-4003. To determine if there are changes in markers (chemicals in the blood) in the blood shown to be related to disease state.

CONTACTS AND LOCATIONS:
Overall Officials: George Tidmarsh, MD, PhD, Study Director
Locations (5):
- United States (5):
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - California Institute of Renal Research, La Mesa, California
  - Denver Nephrology, Denver, Colorado
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - Clinical Advancement Center, PLLC, San Antonio, Texas